CLINICAL TRIAL: NCT03573609
Title: Multicenter, Controlled, Randomized Clinical Trial to Evaluate the Effectiveness and Safety of the New Supratube Invention Device to Prevent Pneumonia Associated With Mechanical Ventilation: " Supra-nav Project "
Brief Title: Evaluation of the Effectiveness and Safety of Supratube Device
Acronym: SUPRANAV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Cardiovascular de Colombia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 0001
Record Dates: First submitted 2018-05-10; First posted 2018-06-29 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2018-04

CONDITIONS: Intensive Critical Unit; Pneumonia; Aspiration; Prevention and Control
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Usual respiratory care
- Supranav (Active Comparator): Respiratory care with "supranav" which is a continuous supraglottic suction device
  Interventions: Device: Supranav

INTERVENTIONS:
Device: Supranav — Continuous supraglottic suction device for patients with orotraqueal intubation an mechanical ventilation
  Arms: Supranav

SUMMARY:
Purpose of the trial:

Trial design: Two-parallel arm, double-blind, individually randomized controlled trial.

Primary endpoint:

Clinical evaluation of sinus, oropharyngeal, tracheal, bronchial or pulmonary infections during orotracheal intubation and hospital admission.

Secondary endpoints:

Volume of oropharyngeal secretions aspirated per unit of time (for 24 hours) by the SupraTube and Complications during the use of the SupraTube device: erosions, lacerations, Bleeding, displacement, migration, need for withdrawal.

Inclusion criteria:

* Adult patient
* Orotracheal intubation ≤ 72 hours
* Hospitalized in ICU
* integrity of upper airways

Exclusion criteria:

* International patients
* Coagulopathic patients
* oncology patients
* patients with maxillofacial surgery
* Absence of close responsible family member
* Tracheostomy, shock, local or systemic non-controlled infection

Trial treatment:

Intervention:

Aspiration of secretions with the supranav device

Control:

Usual respiratory care

Expected sample size, enrollment and expected number of centers:

Sample size = 108

Recruitment start date:

Recruitment end date:

Follow-up end date:

Number of centers: 2

Statistical considerations:

* Intention to treat analysis
* The primary outcomes will be analyzed using

ELIGIBILITY:
Inclusion Criteria:

* Intubated adult patients with mechanical ventilation.
* To have a closest responsible relative
* Integrity of the airways

Exclusion Criteria:

* Need of orofacial, cervical or respiratory tract surgical procedures
* Patients with tracheostomy
* Shock,
* Local or systemic uncontrolled infection
* Blood dyscrasia, neoplastic diseases
* Physiological alteration
* Acute or chronic decompensated pathology that is not controlled at the time of selection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-01-20 (Actual)

PRIMARY OUTCOMES:
Ventilator associated events | 24 hours after extubation
  A group of all the conditions that result in a significant and sustained deterioration in oxygenation, defined as a greater than 20% increase in the daily minimum fraction of inspired oxygen or an increase of at least 3 cm H2O in the daily minimum positive end-expiratory pressure (PEEP) to maintain oxygenation. It is imperative to understand that both infectious conditions (such as tracheitis, tracheobronchitis, and pneumonia) and noninfectious conditions (such as atelectasis, pulmonary embolism, pulmonary edema, ventilator-induced lung injury, and others) may fulfill this VAE definition.

SECONDARY OUTCOMES:
Adverse events | 24 hours after extubation
  Number of patientes with Bleeding and lacerations in the oropharynx

CONTACTS AND LOCATIONS:
Overall Officials: Alba L Ramirez Sarmiento, PhD, Principal Investigator — Fundación Cardiovascular de Colombia
Locations (1):
- Fundación Cardiovascular de Colombia, Piedecuesta, Santander Department, Colombia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Orozco-Levi M, Tiga-Loza DC, Aya O, Reyes CF, Caceres-Rivera D, Espitia A, Rey D, Pedrozo Arias KP, Pizarro C, Sanabria-Barrera SM, Serrano-Diaz N, Castillo VR, Ramirez-Sarmiento A. A Novel Supraglottic Suction Device in Mechanically Ventilated Patients: A Randomized Controlled Trial. Med Devices (Auckl). 2025 Mar 24;18:201-212. doi: 10.2147/MDER.S499924. eCollection 2025. PMID 40161252